CLINICAL TRIAL: NCT01476163
Title: Physician Initiated Expanded Access Request for Treatment Use of Migalastat Hydrochloride (AT1001), an Investigational Treatment for Individual Patients With Fabry Disease (AT1001-188)
Brief Title: Physician Initiated Expanded Access Request for Migalastat in Individual Patients With Fabry Disease
Status: Available | Type: Expanded Access
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: AT1001-188
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-05

CONDITIONS: Fabry Disease
Keywords: AT1001; migalastat; Fabry disease; Fabry; Amicus; lysosomal disease; lysosomal disorder
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate

INTERVENTIONS:
Drug: migalastat HCl 150 mg — 150 mg capsule
  Other Names: AT1001, migalastat
Drug: migalastat HCl 20 mg — 20 mg dispersible tablets; dosing will be based on body weight
  Other Names: AT1001, migalastat

SUMMARY:
This program allows physicians to request permission from Amicus Therapeutics (Amicus) for treatment access to migalastat hydrochloride (HCl) for specific patients with Fabry disease. Treatment is open label.

DETAILED DESCRIPTION:
This Physician Initiated Request program allows physicians to request permission from Amicus to receive migalastat HCl for specific patients with Fabry disease who have a mutation amenable to this treatment, who do not have access to commercial Galafold or available treatment alternatives, or do not meet requirements for participation in an existing migalastat clinical study. Up to 20 patients worldwide may be treated. Patients must meet specific criteria to receive Amicus permission for participation. Key criteria for participation include: At least 2 years old; Confirmed GLA gene mutation shown to be responsive to migalastat; Have no treatment option because either unsuitable for enzyme replacement therapy (ERT) or unable to access ERT.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed GLA mutation predicted to be responsive migalastat in the human embryonic kidney (HEK-293) cell-based assay
* At least 2 years of age
* Strong clinical indication for treatment of Fabry disease
* No other treatment option including either unsuitable for ERT or unable to access ERT
* Appropriate female and male contraception
* Willing to receive treatment with migalastat HCl via this program including having signed an authorization for sharing clinical data

Exclusion Criteria:

* Scheduled for renal or other organ transplant or replacement therapy
* Receiving GLYSET® (miglitol), ZAVESCA® (miglustat) or enzyme replacement therapy FABRAZYME® (agalsidase beta), REPLAGAL™ (agalsidase alpha), or Elfabrio® (pegunigalsidase alfa)
* Contraindication to migalastat, i.e., sensitivity to other iminosugar such as miglustat, miglitol
* Treated with another investigational drug within 30 days of start of migalastat HCl treatment
* Unable to comply with study requirements or deemed otherwise unsuitable for study entry in the opinion of the investigator.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics